CLINICAL TRIAL: NCT05040412
Title: Comparison of the Patients With Diabetes Mellitus Using Either Insulin or Oral Antidiabetic Drug In Terms Of Difficult Laryngoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bagcilar Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Kerem Erkalp, Professor, Bagcilar Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020.01.2.05.015
Record Dates: First submitted 2021-09-02; First posted 2021-09-10 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2021-09

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes mellitus, difficult laryngoscopy, insulin
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: Prospective randomised
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Diabetic mellitus patients using insulin (Experimental): The trachea will be intubated by direct laryngoscopy.
  Interventions: Device: difficult laryngoscopy
- Diabetic patients using oral antidiabetic drug (Experimental): The trachea will be intubated by direct laryngoscopy.
  Interventions: Device: difficult laryngoscopy

INTERVENTIONS:
Device: difficult laryngoscopy — Patients will be intubated with the direct laryngoscope.

SUMMARY:
Diabetes Mellitus is known to be a risk factor for difficult laryngoscopy. Several studies showed that diabetes mellitus is responsible for 30% of difficult laryngoscopy.Insulin and oral antidiabetic drugs are two main current medication prescribed for diabetes patients.Insulin is responsible for muscle hypertrophy and weigh gain.Oral antidiabetic drugs induces muscle atrophy. The aim of this study is to evaluate the differences in the difficult laryngoscopy as a general anesthetic component in patients with Diabetes Mellitus (DM) using either insulin or oral antidiabetic drug (OAD).

DETAILED DESCRIPTION:
DM is accepted as a risk factor for difficult intubation.OAD and insulin are two main pharmacological treatment component of DM.Insulin induces respiratory smooth muscle contraction.Otherwise, OAD drugs ca affect muscle atrophy in patients with type II DM patients.The use of these drugs may affect laryngoscopy during endotracheal intubation,which is a component of general anesthesia.Metformin causes muscle atrophy and weight loss.Some in vitro studies have shown an induction of cell apoptosis with therapeutic doses of sulfonylureas which can lead to atrophy.Glinides can cause atrophy in experimental animals.Hypoglycemia and weight gain are two important side effects of intensive insulin therapy.İnsulin is the major anabolic hormone in the body. Insulin binds to receptors on adipose tissues and potentiate inhibition of lypolysis and storage of triglycerids.And this cause obesity.This is one of the reasons that suggest the relationship between insulin and difficult airway.The effect of insulin on airway smooth muscle leads to increased airway contraction,cell proliferation,and the thicker,stiffer and more hypercontractile airway.In some studies,type II DM patients with duration of more than 5 years switched to insulin therapy and airway hypersensitivity was observed in the first three months.Insulin plays an anabolic role in skeletal muscle by enhancing amino acids transport in skeletal muscle and by increasing the rate of protein synthesis.İnsulin induces air way smooth muscle contraction through the production of contractile prostaglandins, which in turn are dependent on Rho-kinase for their contractile effects.Prostaglandins also stimulate IL-6 and MuRF-1 transcription in human skeletal muscles.Prostaglandin regulates skeletal muscle mass and function.Therefore,insulin may cause airway skeletal muscle contraction and may be the reason of difficult laryngoscopy.

The aim of this study is to evaluate the differences in the difficult laryngoscopy as a general anesthetic component in patients with Diabetes Mellitus (DM) using either insulin or oral antidiabetic drug (OAD).

METHODS After the approval of the local ethics committee of our hospital, a study was planned for a total of 230 patients including Type I and Type II DM patients and non-DM patients as a control group who would undergo elective surgery between 25.01.2020-30.04.2020.Age, gender, body mass index (BMI), Mallampati scores, thyromental distance (TMD), sternomental distance (SMD), inter-incisor distance (ID) and neck extension measurements were taken.Preoperative HbA1C levels, DM type, diagnosis time and duration of insulin or OAD use were recorded.Patients without DM, patients using insulin and patients using OAD were grouped as group C, group I and group D, respectively.DM patients were planned to be operated as first patient in the morning.50 mg of ranitidine,10 mg of metoclopramide and 1 gr of cefazolin for surgical prophylaxis were administered intravenously 30 minutes before anthesia induction.Patients were preoxygenated with 100% O2 for 3 minutes.As diabetes mellitus patients are under high risk of aspiration due to gastroparesis,we applied rapid sequence induction technique.1 mcg/kg fentanyl citrate,2 mg/kg propofol,1mg/kg rocuronium bromide were given intravenously according to patient's adjusted body weight.After low tidal volume ventilation with face mask,the trachea was intubated by using DL (Macintosh laryngoscope).During intubation, the following data were documented:Cormack-Lehane grade, number of laryngoscopic attempts, intubation time, intubation success at the first attempt, performance of backward-upward-rightward pressure (BURP) maneuver and requirement of use of different airway equipments were compared between the groups. Adverse events related to tracheal intubation were evaluated: desaturation (SPO2<94), hypercabia (ETCO2>35), hypertension (mean arterial pressure >20% above baseline values), tachycardia (heart rate >20% above baseline values), new onset arrhythmia, laryngospasm, bronchospasm, airway trauma and sore throat in PACU). The primary outcome measures are mallampati score,thyromental distance,Cormack-Lehane grade and the time to intubation,secondary outcome measures are first-attempt intubation success,number of laryngoscopic attempts,performance of backward-upward-rightward pressure (BURP) maneuver and requirement of use of different airway equipments.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective surgery
* Patients needing endotracheal intubation
* Patients having eithe Type I or Type II diabetes mellitus (those who have been using insulin or OAD for at least the past 5 years)

Exclusion Criteria:

* Emergency surgery
* Difficult intubation story
* İmpaired airway anatomy
* Morbidly obese (BMI > 40 kg/m2)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2020-01-25 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-05-15 (Actual)

PRIMARY OUTCOMES:
Intubation time | 0-120 seconds after intubation.The time elapsed between the passage of the larygoscope through the teeth and the detection of ETCO2
  Mallampati class,Thyromental distance,Cormack Lehane classification,Intubation time

SECONDARY OUTCOMES:
Intubation difficulty | -120 seconds after intubation.The time elapsed between the passage of the larygoscope through the teeth and the detection of ETCO2
  First attempt intubation success rate,numbers of attempt,Application of BURP manauver,number of alternative techniques

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul Bagcilar Egitim ve arastirma hastanesi, Istanbul, Bagcilar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hashim K, Thomas M. Sensitivity of palm print sign in prediction of difficult laryngoscopy in diabetes: A comparison with other airway indices. Indian J Anaesth. 2014 May;58(3):298-302. doi: 10.4103/0019-5049.135042. PMID 25024473
- [Result] Warner ME, Contreras MG, Warner MA, Schroeder DR, Munn SR, Maxson PM. Diabetes mellitus and difficult laryngoscopy in renal and pancreatic transplant patients. Anesth Analg. 1998 Mar;86(3):516-9. doi: 10.1097/00000539-199803000-00012. PMID 9495404
- [Result] Mashour GA, Kheterpal S, Vanaharam V, Shanks A, Wang LY, Sandberg WS, Tremper KK. The extended Mallampati score and a diagnosis of diabetes mellitus are predictors of difficult laryngoscopy in the morbidly obese. Anesth Analg. 2008 Dec;107(6):1919-23. doi: 10.1213/ane.0b013e31818a9946. PMID 19020139
- See also: Dr Priya K et al Sensitivity and Specificity of Palm Print Sign in Difficult Laryngoscopy among Diabetic Patients, JMSCR Volume 06 Issue 09 September 2018 — http://dx.doi.org/10.18535/jmscr/v6i9.127
- See also: Kute R, Gosavi R, Bhaleker P, Phalgune D. Predictability of airway evaluation indices in diabetic and nondiabetic patients requiring general anesthesia with endotracheal intubation. Indian Anaesth Forum 2019;20:70-5 — http://www.theiaforum.org/text.asp?2019/20/2/70/265639